CLINICAL TRIAL: NCT03388359
Title: Role of Extracellular Matrix in the Development of Airway Remodeling in Asthma
Acronym: ECMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Research Council of Lithuania (Other); University of Groningen (Other)
Responsible Party: Principal Investigator, Kestutis Malakauskas, Principal Investigator, Clinical Professor, Head of Laboratory, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P-MIP-17-115; PSUL-010/2014 (Other: Lithuanian University of Health Sciences)
Record Dates: First submitted 2017-08-23; First posted 2018-01-03 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Allergic Asthma; Airway Remodelling; Extracellular Matrix Alteration
Keywords: asthma; eosinophils; Extracellular matrix; airway smooth muscle; airway remodelling; fibroblast
MeSH Terms: conditions — Airway Remodeling; Asthma | interventions — Allergens; Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergic asthma (Experimental): Bronchial asthma and sensitization to D. pteronyssinus allergen Interventions: Bronchial challenge with allergen (Dermatophagoides pteronyssinus, Dosimeter ProvoX (Ganshorns)); Eosinophil and linear bronchial smooth muscle cell or pulmonary fibroblast co-culture formation (eosinophils, fibrobralst, airway smooth muscle cells); Inhibition of Wnt and Smad signaling pathways; Extracellular matrix turnover and deposition assessment.
  Interventions: Procedure: Bronchial challenge with allergen; Other: Co-culture formation; Other: Inhibition of Wnt and Smad signaling pathways; Other: Extracellular matrix turnover and deposition assessment; Biological: Dermatophagoides pteronyssinus allergen; Device: Dosimeter ProvoX (Ganshorn); Biological: Eosinophils; Biological: Airway smooth muscle cells; Biological: Fibroblasts
- Healthy subjects (Active Comparator): Healthy subjects without allergic and other chronic respiratory diseases (control group).
  Interventions: Bronchial challenge with allergen (Dermatophagoides pteronyssinus, Dosimeter ProvoX (Ganshorns)); Eosinophil and linear bronchial smooth muscle cell or pulmonary fibroblast co-culture formation (eosinophils, fibrobralst, airway smooth muscle cells); Inhibition of Wnt and Smad signaling pathways; Extracellular matrix turnover and deposition assessment.
  Interventions: Procedure: Bronchial challenge with allergen; Other: Co-culture formation; Other: Inhibition of Wnt and Smad signaling pathways; Other: Extracellular matrix turnover and deposition assessment; Biological: Dermatophagoides pteronyssinus allergen; Device: Dosimeter ProvoX (Ganshorn); Biological: Eosinophils; Biological: Airway smooth muscle cells; Biological: Fibroblasts

INTERVENTIONS:
Procedure: Bronchial challenge with allergen — Bronchial challenge is performed with D. pteronyssinus allergen. Measurements of differences in eosinophils activity after allergen challenge.
Other: Co-culture formation — Eosinophil and linear bronchial smooth muscle cell or pulmonary fibroblast co-culture formation. Bronchial smooth muscle cell and pulmonary fibroblast proliferation, migration, contractillity, differentiation, eosinophil adhesion to the bronchial smooth muscle cells or pulmonary fibroblast.
Other: Inhibition of Wnt and Smad signaling pathways — Wnt and Smad signaling pathways inhibitors effect on development of airway remodelling processes (extracellular matrix production, bronchial smooth muscle cell and pulmonary fibroblast proliferation, contractillity, differentiation, migration).
Other: Extracellular matrix turnover and deposition assessment — Eosinophils effect on extracellular matrix proteins (collagen, fibronectin, elastin, versican, decorin, laminin, etc.) and matrix metalloproteinasis (MMP-2,9,12,etc.) production by pulmonary fibroblasts.
Biological: Dermatophagoides pteronyssinus allergen — Dermatophagoides pteronyssinus allergen is required to perform allergen bronchial challenge test.
Device: Dosimeter ProvoX (Ganshorn) — Device for allergen bronchial challenge test.
Biological: Eosinophils — Eosinophils are isolated from peripheral blood
Biological: Airway smooth muscle cells — Airway smooth muscle cells from healthy subjects (support from the University of Groningen)
Biological: Fibroblasts — Normal human fibroblast cell lines (commercial fibroblast lines)

SUMMARY:
Asthma is a major noncommunicable chronic inflammatory disorder which is characterized by airway inflammation and related to pathological modifications of the bronchial wall structure so called airway remodeling. Airway remodeling seen in asthma is mainly described by epithelial changes, subepithelial fibrosis, increased airway smooth muscle (ASM) mass, decreased distance between ASM and epithelium, mucous gland and goblet cell hyperplasia, vascular changes and edema. Near these well known pathophysiological changes of the airways, the extracellular matrix (ECM) can be distinguished as a new important factor included in development of airway remodeling in asthma.

DETAILED DESCRIPTION:
Asthma is a major noncommunicable chronic inflammatory disorder which is characterized by airway inflammation and related to pathological modifications of the bronchial wall structure so called airway remodeling. Airway remodeling seen in asthma is mainly described by epithelial changes, subepithelial fibrosis, increased airway smooth muscle (ASM) mass, decreased distance between ASM and epithelium, mucous gland and goblet cell hyperplasia, vascular changes and edema. Near these well known pathophysiological changes of the airways, the extracellular matrix (ECM) can be distinguished as a new important factor included in development of airway remodeling in asthma.

ECM is a building block between airways and lung parenchyma. It plays a crucial role in the maintenance of pulmonary structure and functions influencing the distribution and adhesion of inflammatory cells, fluid balance, elasticity and can act as a resource of inflammatory mediators. In asthma, predominant eosinophilic airway inflammation can result the dysregulation of ECM, which are identified as altered quantitative and qualitative composition of ECM, activated molecular signaling pathways which are responsible for triggered ECM proteins production. The main sources of ECM proteins in lungs are pulmonary fibroblasts and ASM cells. In asthma, fibroblasts are responsive to many inflammatory cytokines which activate and promote fibroblasts proliferation, contractility and cellular differentiation to myofibroblasts form with up-regulated rate of matrix production. In turn, activated fibroblasts secrete cytokines IL-1β, IL-33, CXC, CC chemokines, various types of matrix metalloproteinases (MMPs) as well as reactive oxygen species. These factors allow fibroblasts to assist in the activation and migration of resident immune cells and endow fibroblast roles in chemical and cell-mediated immunity, acute and chronic inflammation, extravasation of immune cells into connective tissue of the lungs. The ASM cells are also the strong contributor to the ECM protein pool in the lungs - they can produce the variety of ECM proteins contributing to the tissue structure and elasticity which are seen unbalanced in asthma. While fibroblasts and ASM cells determine ECM proteins composition, the ECM in turn can affect the structural cells behavior in lung tissue. The role of cell-matrix interactions represents an area for active investigation on the ability of lung matrix to prime the structural pulmonary cells.

The excess of ECM proteins deposition is associated with activation of profibrotic factor transforming growth factor-beta 1 (TGF-β1) mediated WNT and Smad signaling pathways. Highest levels of TGF-β1 in airways are released by eosinophils - the main inflammatory cells in asthma pathogenesis. During stable asthma and especially allergen provoced acute asthma episodes eosinophils infiltrate into the airways, enhancing local levels of TGF-β1 and other various cytokines, chemokines and growth factors near the connective tissue and ASM bundles. However, how eosinophil-released mediators induce ECM dysregulation leading to development of airway remodeling are not investigated part of asthma pathogenesis.

Asthma still cannot be cured, but appropriate management can control the disease severity. Better understanding in development of asthma is the main objective which must to be pursued. Based on this rationale the investigators aimed to investigate eosinophilic airway inflammation mediated production of ECM proteins and MMPs, activity for their release responsible molecular signaling pathways, and how dysregulated ECM affect fibroblasts and ASM cells proliferation, migration, differentiation and contractility in asthma. Trying to understand and control the development of asthma the investigators will use models of combined cells cultures estimating ECM homeostasis in stable and acute asthma. Blocking with specific inhibitors of WNT and Smad signaling pathways, potentially responsible for ECM proteins and MMPs production, will help to find the controlling mechanisms of ECM dysregulation. Therefore, evaluation of ECM proteins degradation fragments and levels of MMPs will help to estimate an applied value of these circulating biomarkers in asthma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18-50 years;
2. Allergic asthma and sensitization to house dust mites (D. pteronyssinus) allergen, approved with:

2. 1. Medical history and symptoms more than one year and 2.2. skin prick test positive for D. pteronyssinus (positive wheals are those exceeding 3mm in diameter greater than the negative control) and 2.3. Positive bronchial challenge with methacholine or documented completely reversible bronchial obstruction; 3. Stable lung function (FEV1≥70 perc.); 4. Postmenopausal women. Premenopausal women if pregnancy test is negative and they agree to use an effective contraceptive measures during the study; 5. Healthy subjects without allergic and other chronic respiratory diseases (control group); 6. Non- smokers; 7. Participants who gave his/her informed written consent.

Exclusion Criteria:

1. Asthma exacerbation 1 month prior to study
2. Clinically significant permanent allergy symptoms (ex. cat or dog dander induced allergy)
3. Contraindications to perform an allergy skin test and/or bronchial provocation test 3.1. Active airway infection 1 month prior the study; 3.2. Used medicaments: 3.2.1. Inhaled glucocorticoids intake 1 month prior the study; 3.2.2. Antihistamines intake 7 days prior the study; 3.2.3. Short acting β2 agonists 12 hours prior the study; 3.2.4. Long acting β2 agonists 2 days prior the study; 3.2.5. Leukotriene receptor antagonists prior 14 days;
4. If the histamine mean wheal diameter is <= 3 mm or control mean wheal diameter is >= 3 mm;
5. Contraindications for epinephrine;
6. Other significant mental and / or internal diseases and conditions, which could be as exclusion criteria due to the opinion of the researcher;
7. Alcohol or narcotic abuse;
8. Pregnancy;
9. Breast-feeding.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-11-10 (Estimated); Study Completion 2020-12-08 (Estimated)

PRIMARY OUTCOMES:
Effect of bronchial challenge with specific allergen on eosinophils activity and impact on pulmonary fibroblasts | First measurements in 24, 48 and 72 h time points after co-culture of eosinophils and pulmonary fibroblasts, summarized data - through study completion, an average of 1 year.
  Bronchial challenge is performed with D. pteronyssinus allergen (HEP/ml). Measurements of altered eosinophils ROS production (changes in pct.), viability (changes in pct.), outer-membrane integrins expression (changes in pct.). Altered fibroblasts apoptosis (changes in pct.), proliferation (changes in pct.), migration (changes in pct.) and contractility (changes in pct.) after co-culture with eosinophils from asthmatic or healthy individuals.
  All mentioned measurements from experimental plan describes one task with final results of increase or decrease in percentage levels.

SECONDARY OUTCOMES:
Extracellular matrix turnover and deposition | First measurement in 24 h time points after co-culture of eosinophils and pulmonary fibroblasts, summarized data - through study completion, an average of 1 year.
  Eosinophils effect on extracellular matrix proteins (collagen, fibronectin, elastin, versican, decorin, laminin, etc.) and matrix metalloproteinasis (MMP-2,9,12,etc.) altered gene expression in folds over control by pulmonary fibroblasts.
  All mentioned measurements from experimental plan describes one task with final results of increase or decrease in folds.
Wnt and Smad signaling pathways inhibitors effect | Through study completion, an average of 1 year.
  Wnt and Smad signaling pathways inhibitors effect on development of airway remodelling processes (changes in pct. of extracellular matrix production, bronchial smooth muscle cell and pulmonary fibroblast proliferation, contractillity, differentiation, migration).
  All selected measurements from experimental plan describes one task with final results of increase or decrease in percentage levels.
Cytokines and growth factors production | Through study completion, an average of 1 year.
  Proinflammatory cytokines and growth factors production (concentration) of eosinophils, bronchial smooth muscle cell and pulmonary fibroblast.
  All selected measurements from experimental plan describes one task with final results of altered concentration (pg/ml; ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Kęstutis Malakauskas, Prof., Dr., Study Chair — Lithuanian University of Health Sciences, Department of Pulmonology
Locations (1):
- Lithuanian University of Health Sciences, Pulmonology Department, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brightling CE, Gupta S, Gonem S, Siddiqui S. Lung damage and airway remodelling in severe asthma. Clin Exp Allergy. 2012 May;42(5):638-49. doi: 10.1111/j.1365-2222.2011.03917.x. Epub 2011 Dec 22. PMID 22192725
- [Background] Januskevicius A, Vaitkiene S, Gosens R, Janulaityte I, Hoppenot D, Sakalauskas R, Malakauskas K. Eosinophils enhance WNT-5a and TGF-beta1 genes expression in airway smooth muscle cells and promote their proliferation by increased extracellular matrix proteins production in asthma. BMC Pulm Med. 2016 Jun 13;16(1):94. doi: 10.1186/s12890-016-0254-9. PMID 27297409
- [Background] Firszt R, Francisco D, Church TD, Thomas JM, Ingram JL, Kraft M. Interleukin-13 induces collagen type-1 expression through matrix metalloproteinase-2 and transforming growth factor-beta1 in airway fibroblasts in asthma. Eur Respir J. 2014 Feb;43(2):464-73. doi: 10.1183/09031936.00068712. Epub 2013 May 16. PMID 23682108
- [Background] Kendall RT, Feghali-Bostwick CA. Fibroblasts in fibrosis: novel roles and mediators. Front Pharmacol. 2014 May 27;5:123. doi: 10.3389/fphar.2014.00123. eCollection 2014. PMID 24904424
- [Background] Amara N, Goven D, Prost F, Muloway R, Crestani B, Boczkowski J. NOX4/NADPH oxidase expression is increased in pulmonary fibroblasts from patients with idiopathic pulmonary fibrosis and mediates TGFbeta1-induced fibroblast differentiation into myofibroblasts. Thorax. 2010 Aug;65(8):733-8. doi: 10.1136/thx.2009.113456. PMID 20685750
- [Background] Bondi CD, Manickam N, Lee DY, Block K, Gorin Y, Abboud HE, Barnes JL. NAD(P)H oxidase mediates TGF-beta1-induced activation of kidney myofibroblasts. J Am Soc Nephrol. 2010 Jan;21(1):93-102. doi: 10.1681/ASN.2009020146. Epub 2009 Nov 19. PMID 19926889
- [Background] Balestrini JL, Chaudhry S, Sarrazy V, Koehler A, Hinz B. The mechanical memory of lung myofibroblasts. Integr Biol (Camb). 2012 Apr;4(4):410-21. doi: 10.1039/c2ib00149g. Epub 2012 Mar 13. PMID 22410748
- [Derived] Janulaityte I, Januskevicius A, Kalinauskaite-Zukauske V, Palacionyte J, Malakauskas K. Asthmatic Eosinophils Promote Contractility and Migration of Airway Smooth Muscle Cells and Pulmonary Fibroblasts In Vitro. Cells. 2021 Jun 4;10(6):1389. doi: 10.3390/cells10061389. PMID 34199925
- [Derived] Kalinauskaite-Zukauske V, Januskevicius A, Janulaityte I, Miliauskas S, Malakauskas K. Serum Levels of Epithelial-Derived Cytokines as Interleukin-25 and Thymic Stromal Lymphopoietin after a Single Dose of Mepolizumab in Patients with Severe Non-Allergic Eosinophilic Asthma: A Short Report. Can Respir J. 2019 Dec 1;2019:8607657. doi: 10.1155/2019/8607657. eCollection 2019. PMID 31885750
- [Derived] Kalinauskaite-Zukauske V, Januskevicius A, Janulaityte I, Miliauskas S, Malakauskas K. Expression of eosinophil beta chain-signaling cytokines receptors, outer-membrane integrins, and type 2 inflammation biomarkers in severe non-allergic eosinophilic asthma. BMC Pulm Med. 2019 Aug 22;19(1):158. doi: 10.1186/s12890-019-0904-9. PMID 31438916